CLINICAL TRIAL: NCT06533228
Title: Comparison of Conventional Clinical and Abbreviated MR Enterography Protocols in Children and Adults With Crohn's Disease
Brief Title: Helmsley 3.0: Abbreviated MRE
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0086
Record Dates: First submitted 2024-07-25; First posted 2024-08-01 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Crohn's Disease
Keywords: Magnetic Resonance Imaging (MRI); Crohn's Disease; Magnetic Resonance Enterography (MRE)
MeSH Terms: conditions — Crohn Disease | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Crohn's Disease Patients: Children and adults, who are scheduled for a clinical magnetic resonance enterography (MRE) to evaluate staging/ restaging of Crohn's disease, will be approached to undergo our novel abbreviated MRE. No intervention, observation only, perform MRE, and complete trade-off tolerance survey.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI) or Magnetic Resonance Enterography (MRE)

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging (MRI) or Magnetic Resonance Enterography (MRE) — Abbreviated magnetic resonance enterography (MRE) imaging to detect active inflammation in patient's with known Crohn's Disease.

SUMMARY:
The purpose of our study is to compare an abbreviated magnetic resonance imaging (MRI) of the bowel or magnetic resonance enterography (MRE) protocol to a conventional, standard of care MRE in children and adults with Crohn's Disease.

DETAILED DESCRIPTION:
This multi-center study will evaluate the effectiveness of an abbreviated magnetic resonance imaging (MRI) of the bowel or magnetic resonance enterography (MRE) to document the presence and severity of small bowel inflammation, the presence and features of stricturing and penetrating disease in children and adults with Crohn's Disease.

The abbreviated MRI of the bowel or MRE will not involve IV contrast or an injection of glucagon and water will replace the oral contrast used in standard of care MREs. Scan time will be greatly reduced with the abbreviated MRE ( approximately 15 minutes) compared to a standard of care MRE (approximately 60 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Established Crohn's disease diagnosis in patients 10 and older
* Undergoing clinical magnetic resonance enterography (MRE) examinations for any reason(s) below

  * Staging/ restaging/ follow- up of intestinal inflammation
  * Evaluation of known or suspected luminal narrowing/ stricturing disease
  * Evaluation of known or suspected internal penetrating disease

Exclusion Criteria:

* Undergoing initial imaging for suspected Crohn's disease where the diagnosis of Crohn's disease has yet to be definitively established
* New Crohn's disease diagnosis, undergoing baseline imaging
* Isolated colonic disease
* Known or suspected pregnancy
* Contraindication to magnetic resonance imaging (MRI)
* Ileostomy or prior ileal resection
* Less than 10 years of age
* Unable or unwilling to follow imaging procedures
* Non- English speaking

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Compare clinical MRE with research MRE | 3 years
  Our abbreviated magnetic resonance enterography (MRE) will be non-inferior to a standard clinical MRE in detecting small bowel inflammation, strictures and penetrating disease associated with Crohn's Disease.

SECONDARY OUTCOMES:
Patient experiences and preferences between the abbreviated MRE and the standard clinical MRE. | 3 years
  Patients/patients parents will answer a survey to determine if the abbreviated magnetic resonance enterography (MRE) or the clinical MRE is preferred.
Willingness to trade diagnostic performance for patient experience | 3 years
  We will ask patients a series of questions to determine their tolerance for trading diagnostic performance for a better patient experience.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Dillman, Principal Investigator — CCHMC
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone, New York, New York

DOCUMENTS (2):
  • Study Protocol (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/28/NCT06533228/Prot_000.pdf
  • Informed Consent Form (2024-06-17): https://cdn.clinicaltrials.gov/large-docs/28/NCT06533228/ICF_001.pdf